CLINICAL TRIAL: NCT07056816
Title: Çocuk Acil Serviste Nebülize İnhalasyon Alan Çocuklarda İnteraktif Oyuncak ve Robot'un Anksiyete ve Korkuya Etkisi: Randomize Kontrollü Çalışma
Brief Title: Effects of Interactive Toys and Robots on Anxiety and Fear in Children Receiving Nebulized Inhalation in the Pediatric Emergency Department
Acronym: social robots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aylin Kurt (Other)
Responsible Party: Sponsor-Investigator, Aylin Kurt, Assistant Professor, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2025-SBB-0315
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-06

CONDITIONS: Child; Fear Anxiety; Inhalant Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive Doll Group (Experimental): Interactive Doll: Their hearts beat and they say "hello" as soon as you put it on your finger because they know it's really yours! They also have a different personality and reactions when they open and close your finger. With sensors in their head, mouth and belly, Fingerlings respond to your touch and will respond to you. You can also shake them and turn them upside down for even more reactions because they love to monkey around. And their positive tail can hang down or flip up so they can sit on your table or shelf. Kids will play with the Interactive Doll during the inhalation treatment.
  Interventions: Other: Interactive Doll
- Interactive Robot Group (Experimental): Interactive Robot: It has an interactive design that improves children's music listening and learning skills. It attracts children's attention with its vibrant colors and cute design, and teaches them while having fun. It has a voice imitation feature and a response feature that makes different sounds when its head is touched. Children will play with the Interactive Robot during inhalation treatment.
  Interventions: Other: Interactive Robot
- Control Group (No Intervention): The standard information given to all children receiving nebulized inhalation treatment in the pediatric emergency department will be given to the children in the control group.

INTERVENTIONS:
Other: Interactive Doll — Interactive Doll: Their hearts beat and they say "hello" as soon as you put it on your finger because they know it's really yours! They also have a different personality and reactions when they open and close your finger. With sensors in their head, mouth and belly, Fingerlings respond to your touch and will respond to you. You can also shake them and turn them upside down for even more reactions because they love to monkey around. And their positive tail can hang down or flip up so they can sit on your table or shelf. Kids will play with the Interactive Doll during the inhalation treatment.
  Arms: Interactive Doll Group
Other: Interactive Robot — Interactive Robot: It has an interactive design that improves children's music listening and learning skills. It attracts children's attention with its vibrant colors and cute design, and teaches them while having fun. It has a voice imitation feature and a response feature that makes different sounds when its head is touched. Children will play with the Interactive Robot during inhalation treatment.
  Arms: Interactive Robot Group

SUMMARY:
Pediatric emergency services are of critical importance for pediatric patients admitted due to sudden illnesses and traumas. However, these environments are serious sources of stress and anxiety for children due to reasons such as uncertainty, pain, and separation anxiety. The emergency service experience can have long-term effects on the child's psychological state and negatively affect the success of medical interventions. Therefore, the development and implementation of various methods to reduce children's anxiety has become a great necessity. In recent years, interactive toys and robotic systems have been increasingly used in medical settings to reduce children's anxiety. Such technological tools have been shown to provide emotional support to children, reduce stress levels by distracting them, and make medical procedures more tolerable. However, there is not enough evidence-based research on the effectiveness of interactive toys and robots, especially in emergency settings, during common but frightening procedures such as nebulized inhalation. This study aims to evaluate the effect of interactive toys and robots on anxiety and fear in children receiving nebulized inhalation treatment in pediatric emergency services. This study, which will be conducted using a randomized controlled design, will make a significant contribution to understanding and improving children's psychological responses to medical procedures. The study was planned as a randomized controlled trial. The population of this study will be conducted in the pediatric emergency department of Ankara Provincial Health Directorate Yıldırım Beyazıt University Yenimahalle Education and Research Hospital between 05.05.2025-05.05.2026. The sample of this study will consist of 72 children aged between 4-10 who agreed to participate in the study and met the inclusion criteria and who received nebulized inhalation treatment and met the inclusion criteria.

Hypotheses of the study:

H0 = Playing with interactive toys and interactive robots during nebulized inhalation treatment has no effect on anxiety and fear in children.

H1 = Playing with interactive toys and interactive robots during nebulized inhalation treatment is effective in reducing anxiety and fear in children.

ELIGIBILITY:
Inclusion Criteria:

* Being a child between the ages of 4-10,
* Receiving nebulized inhalation treatment in the pediatric emergency department,
* The parent agreeing to participate in the research,
* The child not having speech or vision impairments or any other disabilities that would hinder or prevent communication.

Exclusion Criteria:

* Children whose parents' permission cannot be obtained
* The child's speech and vision impairment, or any other disability that would make communication difficult or prevent it.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
The level of anxiety is evaluated using the Children Anxiety Meter-State | during the procedure
  The Children's Anxiety Meter (CAM-S) assesses children's anxiety in clinical settings and is used prior to medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom and contains horizontal lines at intervals going upwards. Scale scores range from 0 to 10, where higher values represent higher anxiety. Personal reports and records from children, their parents, the researcher, and the nurse, who are asked to mark the scale with a pen, are used to assess the anxiety levels of children

SECONDARY OUTCOMES:
The level of anxiety is evaluated using the Child Fear Scale | during the procedure
  Child Fear Scale assesses children's fear in clinical settings and is used prior to medical procedures. The Child Fear Scale (CFS) consists of facial expressions ranging from a neutral face on the far left (0 points: no fear/anxiety) to a frightened face on the far right (4 points: extreme fear/anxiety). Children are asked to mark their level of fear or anxiety by choosing the most appropriate facial expression to represent them. Personal reports and records from children, their parents, the researcher, and the nurse, who are asked to mark the scale with a pen, are used to assess the anxiety levels of children.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol